CLINICAL TRIAL: NCT06828224
Title: Open, Non-comparative Study to Evaluate the Effectiveness and Safety of the Medical Device KOS® L in Correcting Moderate or Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Beauty Kozmetik (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGMQUA/0324/MD
Record Dates: First submitted 2025-02-05; First posted 2025-02-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-06

CONDITIONS: Nasolabial Fold
Keywords: "Moderate" or "Severe" nasolabial folds (NLFs)
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOS® L (Other): An open, non-comparative, interventional single-armed clinical trial.
  Interventions: Device: KOS® L

INTERVENTIONS:
Device: KOS® L — Delivery of medical device as injection

SUMMARY:
The utilization of minimally invasive techniques has brought about a transformative shift in the approach to face rejuvenation, potentially representing one of the most notable advancements in facial plastic surgery in recent times. Originally employed to address the presence of fine lines and wrinkles, the application of fillers has now evolved to encompass the remediation of volume depletion and the enhancement of the aging visage.

KOS® L in the dermis regulates water balance, osmotic pressure and ion flow and functions as a sieve, excluding certain molecules, enhancing the extracellular domain of cell surfaces and stabilizes skin structures by electrostatic interactions.

The Research Question of the present study is the following: to collect sufficient clinical data to demonstrate compliance with the General Safety and Performance Requirements of KOS® L when used as intended.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the subject
* Men and women with ≥ 22 years of age
* Two fully visible bilateral nasolabial folds, each with a Wrinkle Severity Rating Scale Score of moderate (3) or severe (4) based on the 5-point WSRS
* Ability to follow study instructions and likely to complete all required visits
* Reliable methods of contraception which result in a low failure rate (i.e. less than 1 % per year) for women of childbearing potential, e.g. implants, injectables, combined oral contraceptives, some intrauterine-devices, sexual abstinence or vasectomized partner) for the entire study duration.

Exclusion Criteria:

1. Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable permanent filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …)
2. Subject who received oral surgery (e.g. tooth extraction, orthodontia or implantation) within 6 weeks prior to screening visit or who plans to undergo any of these procedures during the study
3. Severe midface volume loss or severity of wrinkles or folds requiring other treatments
4. Previous tissue revitalization with neurotoxin, laser or light, mesotherapy, chemical peeling, or dermabrasion below the zygomatic arch within 6 months
5. Previous tissue augmenting therapy or, contouring, or fat injection in the facial area
6. Subject with a tattoo, a scar, moles or anything on the studied zones which might interfere with the evaluation
7. Subject having received injection with a resorbable filling product (eg, hyaluronic acid, collagen) below the inferior orbital rim within the past 12 months prior to screening visit
8. History of allergy to lidocaine or local anaesthesia of amide compounds
9. Suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…)
10. Body mass index BMI<18 or >30 kg/m2
11. Smoker with >10 pack-year history within the past year
12. Using any new over-the-counter or prescription oral or topical, anti-wrinkle products within 30 days before enrolment or is planning to begin using such products during the study. (Subjects who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study)
13. History of or active autoimmune disease/immune deficiency
14. Prone to hypertrophic scars
15. History of allergy to hyaluronic acid or any of the product's components
16. Known case of porphyria
17. Pregnancy or lactation
18. Taking medications and/or substances known to increase coagulation time (e.g., aspirin, ibuprofen, or herbal supplements) 10 days prior to treatment
19. Have a condition or be in a situation that, in the physician's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
20. Untreated epilepsy
21. Hypersensitivity to gram positive bacterial proteins as hyaluronic acid is produced by Streptococcus type bacteria.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with at least 1-point improvement from baseline on the WSRS | 6 month
  Proportion of subjects with at least 1-point improvement from baseline on the WSRS (Wrinkle Severity Rating Scale) at month 6 after the last treatment (response rate).
  Wrinkle Severity Rating Scale - from 1 (No visible nasolabial folds) to 5 (Extremely long and deep nasolabial folds)

SECONDARY OUTCOMES:
Change in Wrinkle Severity Rating Scale from baseline | 1, 3, 6 and 12 months
  Change in WSRS (Wrinkle Severity Rating Scale) from baseline at 1, 3, 6 and 12 months after the last treatment.
  Wrinkle Severity Rating Scale - from 1 (No visible nasolabial folds) to 5 (Extremely long and deep nasolabial folds)
Proportion of participants with at least 1-point improvement from baseline on the WSRS | 1, 3 and 12 months
  Proportion of participants with at least 1-point improvement from baseline on the WSRS (Wrinkle Severity Rating Scale) at 1, 3 and 12 months after the last treatment (response rates) Wrinkle Severity Rating Scale - from 1 (No visible nasolabial folds) to 5 (Extremely long and deep nasolabial folds)
Change from baseline in FACE-Q Satisfaction with Facial Appearance | 1, 3, 6 and 12 months
  Change from baseline in FACE-Q Satisfaction with Facial Appearance at 1, 3, 6 and 12 months after the last treatment FACE-Q Satisfaction with Facial Appearance scale - from 1 (Very Dissatisfied) to 4 (Very satisfied)
Proportion of participants having a positive aesthetic evolution on the 5-point GAIS | 1, 3, 6 and 12 months
  Proportion of participants having a positive aesthetic evolution on the 5-point Global Aesthetic Improvement Scale (GAIS) evaluated by the physician and subject at 1, 3, 6 and 12 months after the last treatment.
  5-point Global Aesthetic Improvement Scale - from 1 (very much improved) to 5 (worse)
Short- and long-term adverse effects | 6 and 12 months
  Short- and long-term adverse effects within 2 weeks of the initial or touch-up treatment and during 6, 12 months after the last treatment of the study course, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Behnam D Bayatani, Study Chair
Locations (1):
- Clinica Beyond Dental, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attenello NH, Maas CS. Injectable fillers: review of material and properties. Facial Plast Surg. 2015 Feb;31(1):29-34. doi: 10.1055/s-0035-1544924. Epub 2015 Mar 12. PMID 25763894
- [Background] Monheit G, Beer K, Hardas B, Grimes PE, Weichman BM, Lin V, Murphy DK. Safety and Effectiveness of the Hyaluronic Acid Dermal Filler VYC-17.5L for Nasolabial Folds: Results of a Randomized, Controlled Study. Dermatol Surg. 2018 May;44(5):670-678. doi: 10.1097/DSS.0000000000001529. PMID 29701621
- See also: Champely, S. (2020). pwr: Basic Functions for Power Analysis. R package version 1.3-0. — https://CRAN.R-project.org/package=pwr